CLINICAL TRIAL: NCT04776265
Title: Real World Evidence of Brentuximab Vedotin Consolidation in Patients With Relapsed/Refractory Classical Hodgkin Lymphoma Who Receive Salvage Chemotherapy and Autologous Stem Cell Transplant
Brief Title: RWE of Brentuximab Vedotin Consolidation in Patients With RR HL Who Receive Salvage Chemotherapy and ASCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grupo Argentino de Tratamiento de la Leucemia Aguda (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: GATLA RR-HL-2020
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Hodgkin Lymphoma, Adult; Relapsed Hodgkin's Disease, Adult; Refractory Hodgkin Lymphoma
Keywords: Relapsed/ Refractory Hodgkin Lymphoma; Autologous Stem Cell Transplant; Consolidation; Brentuximab Vedotin
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RR HL Who Receive Salvage Chemotherapy and ASCT: Patients With Relapsed/Refractory Classical Hodgkin Lymphoma Who Receive Salvage Chemotherapy and Autologous Stem Cell Transplant
  Interventions: Other: Evaluation of therapeutical approach after ASCT

INTERVENTIONS:
Other: Evaluation of therapeutical approach after ASCT — Evaluation of therapeutical approach after ASCT

SUMMARY:
This is a multicenter, observational real world study with prospective follow up that will evaluate the treatment approach in patients with relapsed/refractory cHL who undergo ASCT in Argentina.

DETAILED DESCRIPTION:
The purpose of the study is to gather real world evidence of the proportion and characteristics of patients with relapsed refractory cHL who undergo ASCT, who receive consolidation with BV, and to study the factors that determine BV consolidation after ASCT in real world setting.

This study will evaluate the treatment approach in patients with relapsed/refractory cHL who undergo ASCT. All consecutive adult patients with relapsed/refractory cHL who undergo ASCT, regardless of the prior indication to receive or not BV consolidation therapy, will be included in this study and prospectively followed according to local practice.

Patients will be treated and monitored by their physicians according to local clinical practice and guided by the local approved label for patients receiving BV consolidation. Usual follow-up will be determined by the treating physicians' standards of care, and no scheduled patient visits are required for the conduct of this study. There are no visits or specific procedures planned by protocol, however, baseline and follow up data will be gathered every time the patient's response to treatment is assessed or has a medically important event.

All patients that undergo ASCT will be included in final analysis of the primary objectives (Full study population). Patients that receive BV consolidation or not (Non-BV consolidation) will be included in the analysis.

Patients included in the study are expected to be recruited during 24 months and followed up to progression, death, lost to follow or end of study (12 months after the inclusion of the last patient), whatever occurs earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.
* All patients with histologically confirmed cHL who are primary refractory or relapse and receive ASCT as part of their salvage therapy.
* Signature of the form consent for participation in the study.

Exclusion Criteria:

* Patients with Relapsed/Refractory cHL not suitable for ASCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with relapsed/ refractory HL who receive ASCT from main transplant centers in Argentina
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate proportion of patients who received Brentuximab Vedotin and ASCT. | 24 months
  Study real world evidence of the proportion and characteristics of patients with relapsed refractory cHLwho undergo ASCT, who receive consolidation with BV.
Evaluate factors that determine BV consolidation after ASCT. | 24 months
  Study the factors that determine BV consolidation after ASCT in real world setting.

SECONDARY OUTCOMES:
PFS of the whole patient population. | 24 months
OS of the whole patient population. | 24 months
PFS of patients after ASCT who receive consolidation with BV. | 24 months
OS of patients after ASCT who receive consolidation with BV. | 24 months
PFS of patients after ASCT who do not receive consolidation with BV. | 24 months
OS of patients after ASCT who do not receive consolidation with BV. | 24 months
PFS according to PET status at time of ASCT, and other risk factors in patients who receive BV consolidation. | 24 months
OS according to PET status at time of ASCT, and other risk factors in patients who receive BV consolidation. | 24 months
Incidence of Treatment-Emergent Adverse Events of BV consolidation therapy. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Fiad, Principal Investigator — Grupo Argentino de Tratamiento de la Leucemia Aguda; Florencia Negri Aranguren, Principal Investigator — Grupo Argentino de Tratamiento de la Leucemia Aguda
Locations (15):
- Argentina (15):
  - Hospital Nacional Posadas, El Palomar, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Hospital de Alta Complejidad El Cruce, San Juan Bautista, Buenos Aires
  - Hospital San Martín, Paraná, Entre Ríos Province
  - Instituto Privado de Hematologia y Hemoterapia, Paraná, Entre Ríos Province
  - Hospital Escuela de Agudos Dr. Ramón Madariaga, Posadas, Misiones Province
  - IDHEA Clínica Hematológica, Rosario, Santa Fe Province
  - CEMIC, CABA
  - FLEMING, CABA
  - FUNDALEU, CABA
  - Hospital Alemán, CABA
  - Instituto de Trasplantes de Alta Complejidad, CABA
  - Sanatorio Anchorena, CABA
  - Clínica Universitaria Reina Fabiola, Córdoba
  - Hospital Privado de Córdoba, Córdoba

IPD SHARING:
Plan to Share IPD: Yes
Share study protocol
Supporting Information: Study Protocol
Time Frame: The data will become available on May 2021, and will remain available until the end of the clinical trial.